CLINICAL TRIAL: NCT07270432
Title: Randomized Clinical Trial to Evaluate the Safety and Efficacy of Product DNN.65.21.005 in Alleviating Lower Urinary Tract Symptoms in Patients With Benign Prostatic Hyperplasia
Brief Title: Efficacy/ Safety of Product DNN.65.21.005 in Patients With Benign Prostatic Hyperplasia
Acronym: NICCOLO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACH-DTS-03(03/22)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Hyperplasia, Benign
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product DNN.65.21.005 (Experimental)
  Interventions: Drug: Product DNN.65.21.005
- Combodart® (Active Comparator)
  Interventions: Drug: Combodart®

INTERVENTIONS:
Drug: Product DNN.65.21.005 — One capsule every 24 hours
  Arms: Product DNN.65.21.005
Drug: Combodart® — One capsule every 24 hours
  Arms: Combodart®

SUMMARY:
To evaluate the safety and efficacy of DNN.65.21.005 versus Combodart® in the treatment of benign prostatic hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged 50 years and older.
* Ability to understand the study and provide informed consent, documented by signing the Informed Consent Form (ICF).
* Participants presenting lower urinary tract symptoms (LUTS) associated with prostate enlargement, without neurological or infectious causes.

Exclusion Criteria:

* History or evidence of prostate cancer.
* Urinary retention ≥100 mL, as assessed by abdominal prostate ultrasound.
* Previous diagnosis of Parkinson's disease or other neurological disorders that may lead to neurogenic bladder.
* Use of herbal treatments for prostate enlargement within 14 days prior to the screening visit.
* Current use or use of alpha-blocker medications within 7 days prior to the start of study treatment.
* Current use or use of 5-alpha reductase inhibitors (5ARIs) within 180 days prior to the start of study treatment.
* Use of any prohibited medications within the timeframe specified in the study protocol.
* Any clinical findings or observations (clinical or physical evaluation) that, in the investigator's judgment, pose a risk to participation in the study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | 180 days
  Change in International Prostate Symptom Score (IPSS) evaluated 180 days after starting treatment compared to the baseline